CLINICAL TRIAL: NCT02927054
Title: Effect of Education on Resident Physician Knowledge of Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00075424
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Internal Medicine Residents (Other): Sepsis education provided to internal medicine residents
  Interventions: Other: Sepsis Education
- Emergency Medicine Residents (Other): Sepsis education provided to emergency medicine residents
  Interventions: Other: Sepsis Education
- Orthopedic Residents (Other): Sepsis education provided to orthopedic residents
  Interventions: Other: Sepsis Education
- Neurosurgery Residents (Other): Sepsis education provided to neurosurgery residents
  Interventions: Other: Sepsis Education
- General Surgery Residents (Other): Sepsis education provided to general surgery residents
  Interventions: Other: Sepsis Education

INTERVENTIONS:
Other: Sepsis Education — Education provided to hospital residents for the recognition and treatment of systemic inflammatory response syndrome (SIRS), sepsis and severe sepsis

SUMMARY:
A questionnaire was provided, including clinical vignettes and free text answers, to assess and evaluate the ability of resident physicians to identify systemic inflammatory response syndrome (SIRS), sepsis, and severe sepsis. Questionnaire scores were compared between specialties. A whole-hospital educational campaign was provided with the aim to improve sepsis recognition, and the questionnaire survey was repeated after one year to assess the effect of the education on the recognition of sepsis.

DETAILED DESCRIPTION:
Sepsis is the number one cause of mortality in US hospitals. An aim of this study was to evaluate the ability of resident physicians with different training backgrounds to recognize SIRS, sepsis, and severe sepsis. A survey assessment of the definition of SIRS, sepsis, and severe sepsis was administered to internal medicine, emergency room, orthopedic, neurosurgery, and general surgery residents. Then, an intensive educational campaign designed to improve recognition of the patient with sepsis was launched. For approximately 1 year, posters with this educational information were displayed in the hospital, one-on-one educational sessions were provided to residents, and didactic sessions focusing on sepsis were conducted. The survey was then redesigned and administered it to the same groups as described previously.

ELIGIBILITY:
Inclusion Criteria:

Resident physician in an University of Utah training program

Exclusion Criteria:

Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in sepsis recognition and treatment survey score | Baseline and 1 Year
  Questionnaire scores assessing sepsis recognition and treatment at baseline compared to a similar survey following one year of whole-hospital educational campaign, across groups of residents of different training backgrounds

CONTACTS AND LOCATIONS:
Overall Officials: Devin J Horton, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: Yes
If requested, will share with other authors or institutions

REFERENCES:
- [Background] Poeze M, Ramsay G, Gerlach H, Rubulotta F, Levy M. An international sepsis survey: a study of doctors' knowledge and perception about sepsis. Crit Care. 2004 Dec;8(6):R409-13. doi: 10.1186/cc2959. Epub 2004 Oct 14. PMID 15566585
- [Result] Assuncao M, Akamine N, Cardoso GS, Mello PV, Teles JM, Nunes AL, Maia MO, Rea-Neto A, Machado FR; SEPSES Study Group. Survey on physicians' knowledge of sepsis: do they recognize it promptly? J Crit Care. 2010 Dec;25(4):545-52. doi: 10.1016/j.jcrc.2010.03.012. Epub 2010 Jun 19. PMID 20646902